CLINICAL TRIAL: NCT06408012
Title: Enabling Neuroscience Research Approaches for Brain, feeLings and Emotions (ENABLE): An Innovative Platform for Clinical Trials in Mood Disorders
Brief Title: An Innovative Master Platform for Clinical Trials in Mood Disorders
Acronym: ENABLE
Status: Recruiting | Type: Observational
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: Unity Health Toronto (Other); Centre for Addiction and Mental Health (Other); Queen's University (Other); University of Ottawa (Other); University of British Columbia (Other); University of Calgary (Other); McGill University (Other); Nova Scotia Health Authority (Other); University of Michigan (Other); Simon Fraser University (Other); University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Benicio Frey, Professor, Department of Psychiatry and Behavioural Neurosciences, St. Joseph's Healthcare Hamilton
Other Study IDs: CAN-BIND-18
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Mood Disorders; Depressive Disorder; Bipolar and Related Disorders
MeSH Terms: conditions — Mood Disorders; Depressive Disorder; Bipolar and Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Blood Plasma: Venous blood will be collected in blood collection tubes, followed by centrifugation in a refrigerated centrifuge to obtain the plasma. The entire plasma sample from each tube will be equally divided into labelled cryovials (each minimum 1 mL) and stored at -80oC at the clinical site.
  Peripheral Blood Mononuclear Cells (PBMCs): Venous blood will be collected in blood collection tubes, followed by centrifugation and processing to obtain PBMCs that will be divided in 1 ml labeled aliquots and stored at -80oC at the clinical site.
  Whole blood for RNA analysis: Venous blood will be collected in blood collection tubes, processed following the most updated SOP, labeled, and stored at -80oC at each clinical site.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Mood disorders such as depression and bipolar disorder affect over 350 million people around the world. While several effective treatments exist, it is often difficult to match the right treatment to an individual person. Repeated efforts to find the right treatment contribute to poor functioning, low quality of life, and prolongs the time it takes to get well. Most areas of medicine are able to use 'biomarkers' or clinical tests, blood tests, or imaging to help diagnose and treat illness. The search for biomarkers in mood disorders is advancing, but one roadblock to progress is the lack of large, standardized studies of mood disorders that are needed to accurately identify biomarkers. The aim of the ENABLE platform is to provide the Canadian neuroscience community a standardized way of collecting biomarker data from individuals with a range of mood disorders symptoms. In addition, this 'master clinical trial platform' framework will provide a pool of participants who can be recruited into biomarker-based clinical trials.

DETAILED DESCRIPTION:
The ENABLE platform offers to the Canadian neuroscience community (1) standardized data collection methods with deep clinical and neurobiological phenotyping of individuals across the spectrum of mood disorder symptoms; (2) a recruitment pool for efficient launch of clinical trials; and (3) an open source of clinical and neurobiological data for discovery analyses and/or grant applications.

The assessments have been categorized into a tiered system, where participants must consent to complete tier 1 items in order to be enrolled in the platform. Tier 2 items will be optional measures, the absence of these measures will not compromise the inclusion in the platform. A separate written informed consent to be contacted regarding participation in future clinical trials associate with the ENABLE platform will also be offered.

At tier 1, individuals complete clinical assessments (clinician administered and self-report) and during their tier 2, they provide blood, undergo neuroimaging procedures (MRI and EEG); and are given an actigraphy device to wear for two weeks.

ELIGIBILITY:
Inclusion Criteria

Patients:

1. 16 years of age or older.
2. Meet criteria for bipolar or depressive disorders as defined by DSM-5.
3. Fluency in English, sufficient to complete the interviews and self-report questionnaires.

Inclusion Criteria

Healthy Comparison (HC) Participants:

1. 16 years of age or older.
2. No history of psychiatric disorders (according to DSM-5) or significant unstable medical conditions.
3. Fluency in English, sufficient to complete the interviews and self-report questionnaires.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals who meet criteria for bipolar or depressive disorders as defined by DSM-5.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2023-10-17 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Rate of participation in the master trial platform | 31st March 2026
  Number of participants who consent to be included in the registry

CONTACTS AND LOCATIONS:
Overall Officials: Benicio N Frey, Principal Investigator — St. Joseph's Healthcare Hamilton
Locations (9):
- Canada (9):
  - University of Calgary, Calgary, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - McMaster University, Hamilton, Ontario
  - Queen's University, Kingston, Ontario
  - University of Ottawa, Ottawa, Ontario
  - University Health Network, Toronto, Ontario
  - Centre for Addiction and Mental Health, Toronto, Ontario
  - Ontario Shores Centre for Mental Health Sciences, Whitby, Ontario

IPD SHARING:
Plan to Share IPD: Yes
This study is funded by the Ontario Brain Institute (OBI) and Brain Canada. Data collected from this study is entered into a research database called "Brain-CODE",(https://www.braincode.ca/content/about-brain-code), which is currently hosted on high performance computing nodes at the Centre for Advanced Computing (CAC) (https://cac.queensu.ca/) at Queen's University in Ontario, Canada. Participant data will be available to the neuroscience community. Through Brain-CODE, data can be available by submitting a secure form which will need to be done across all platform sites in order to access the data. The IPD that will be shared could include clinical assessments (clinician administered and self-report), neuroimaging (EEG and MRI), and actigraphy data.
Supporting Information: Study Protocol
Time Frame: Currently till the end of March, 2026.
Access Criteria: By application.
URL: https://braininstitute.ca/research-data-sharing/depression